CLINICAL TRIAL: NCT05184673
Title: Moderate Aerobic Activity Through Yoga
Acronym: MAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Samantha M Harden, Principal Investigator, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 21-325
Record Dates: First submitted 2021-08-26; First posted 2022-01-11 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Physical Activity
Keywords: yoga; heart rate; exercise
MeSH Terms: conditions — Motor Activity | interventions — Environment

STUDY DESIGN:
Intervention Model Description: Each group of participants will complete four different yoga classes - hatha thermo-neutral, flow thermo-neutral, hatha hot, and flow hot - in different orders, keeping the time of the class, the other participants in the class, the instructor, and the sequence of the moves the same.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- hatha thermo-neutral (Active Comparator): The hatha classes will hold each pose for 5 breaths in a room temperature (~70 degrees Fahrenheit) space. Yoga sessions will be led by a 500hr Registered Yoga Teacher. This reduces the risk for injury due to the extensive training the yoga teacher will have received and the knowledge of cuing and sequencing for best practice. All study personnel will be vaccinated against SARS-CoV-2, reducing the risk of spreading SARS-CoV-2.
  Interventions: Other: Behavioral and environmental
- hatha hot (Active Comparator): The hatha hot classes will hold each pose for 5 breaths in a room heated to 95 degrees Fahrenheit. Yoga sessions will be led by a 500hr Registered Yoga Teacher. This reduces the risk for injury due to the extensive training the yoga teacher will have received and the knowledge of cuing and sequencing for best practice. All study personnel will be vaccinated against SARS-CoV-2, reducing the risk of spreading SARS-CoV-2.
  Interventions: Other: Behavioral and environmental
- flow thermo-neutral (Active Comparator): The flow hot classes will flow from each pose (one breath per movement) a room temperature (~70 degrees Fahrenheit) space. Yoga sessions will be led by a 500hr Registered Yoga Teacher. This reduces the risk for injury due to the extensive training the yoga teacher will have received and the knowledge of cuing and sequencing for best practice. All study personnel will be vaccinated against SARS-CoV-2, reducing the risk of spreading SARS-CoV-2.
  Interventions: Other: Behavioral and environmental
- flow hot (Active Comparator): The flow hot classes will flow from each pose (one breath per movement) in a room heated to 95 degrees Fahrenheit. Yoga sessions will be led by a 500hr Registered Yoga Teacher. This reduces the risk for injury due to the extensive training the yoga teacher will have received and the knowledge of cuing and sequencing for best practice. All study personnel will be vaccinated against SARS-CoV-2, reducing the risk of spreading SARS-CoV-2.
  Interventions: Other: Behavioral and environmental

INTERVENTIONS:
Other: Behavioral and environmental — These are all active comparator yoga sequences

SUMMARY:
The 2018 Physical Activity Guidelines for Americans (PAGA) recommend 150 minutes of moderate intensity activity for adult (18 years and older) Americans to promote health. PAGA also recommends that older adults (65+) engage in multicomponent and balance exercises weekly as a way to reduce falls and injuries from falls. This recommendation includes yoga, however, the current research and recommendations on using yoga to meet moderate intensity activity guidelines is limited. This study will utilize heart rate monitoring to determine if certain styles of yoga can be used to meet the PAGA.

DETAILED DESCRIPTION:
The 2018 Physical Activity Guidelines for Americans recommend 150 minutes of moderate intensity physical activity each week to promote health. The most recent scientific advisory committee had insufficient evidence to provide recommendations on how the physical practice of yoga fits into the physical activity guidelines. Currently, there have been few studies done on yoga and its relative intensity. Previous randomized, cross-over trial to determine the effects of room temperature (hot yoga versus thermo-neutral environment) on subjective and objective markers of exercise intensity. They concluded that using objective markers (%VO2max) both thermo-neutral and hot yoga would be considered light intensity activity. Previous investigation of power yoga, heart rate, skin temperature, and body mass to determine that power yoga could be considered a moderate-vigorous intensity activity.

Currently, there is a gap in the research on understanding the intensity of exercise offered within a typical yoga studio including "flow", hatha/classical, and hot yoga. Most yoga classes are about 60 minutes in length, and yoga classes of that length have not been investigated. There is also minimal research done on whether wearable activity trackers and accelerometers are able to accurately assess heart rate, and therefore activity intensity level in a yoga setting.

ELIGIBILITY:
Inclusion Criteria:

* Assessed as physical activity readiness i. For those 65-70 years of age. We will also use the Physical Readiness Questionnaire Plus-this "plus" version was developed to be more inclusive of those with limited mobility and not to over-exclude older adults in other clinical trials. If a participant fails the Physical Activity Readiness Questionnaire + (PARQ+), a physician's approval will be mandatory ii. For those 70-85 years of age. Complete PARQ+ as well as physician approval.
* Comprehension of English language
* Able to physically attend class at the yoga studio

Exclusion Criteria:

* Contraindication to physical activity including but not limited to people who can independently walk and stand. This will be part of the verbal screening protocol using Falls Efficacy Scale (FES). This scale has a minimum of 16 (no concern about falling) to maximum of 64 (severe concern about falling). Participants with FES score > 23 will be deemed high concern about falling and be excluded from participation.
* Assesses the presence and severity of 13 psychiatric symptom domains that cut across diagnostic boundaries. These domains include depression, anger, mania, anxiety, somatic symptoms, sleep disturbance, psychosis, obsessive thoughts and behaviors, suicidal thoughts and behaviors, substance use (e.g., alcohol, nicotine, prescription medication, and illicit substance use), personality functioning, dissociation, and cognition/memory problems in adults. Level 1 of this measure includes 23 questions across the 13 domains.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2021-10-28 (Actual)

PRIMARY OUTCOMES:
Continuous heart rate | orientation to week 0 (baseline)
  Polar Version OH1
Continuous heart rate | orientation to week 1
  Polar Version OH1
Continuous heart rate | orientation to week 1.5
  Polar Version OH1
Continuous heart rate | orientation to week 2
  Polar Version OH1
Continuous heart rate | orientation to week 2.5
  Polar Version OH1

SECONDARY OUTCOMES:
Modified Borg Scale | orientation to week 1
  2-items, 1 (very light activity) -10 (maximal effort)
Modified Borg Scale | orientation to week 1.5
  2-items, 1 (very light activity) -10 (maximal effort)
Modified Borg Scale | orientation to week 2
  2-items, 1 (very light activity) -10 (maximal effort)
Modified Borg Scale | orientation to week 2.5
  2-items, 1 (very light activity) -10 (maximal effort)
Yoga Self Efficacy Scale | Baseline
  12-item, 9 point Likert scale, higher score, more self-efficacious
Stanford Leisure-Time Activity Categorical Item | Baseline
  Score of 1-6, higher is better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Samantha M Harden, PhD, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (1):
- Samantha M Harden, Blacksburg, Virginia, United States

IPD SHARING:
Plan to Share IPD: No